CLINICAL TRIAL: NCT05578924
Title: Factors Associated With Gynecological Consultation by General Practitioner
Acronym: Gyn-MG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_008_Gyn-MG
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Adult Daughters
Keywords: Adult women; gynecological acts; general practitioners

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: " women group " — women aged more than 18 years old

SUMMARY:
Because of the shortage of doctors in France, notably gynaecologist, general practitioners are definitely an essential partner women's health. However, few of them regularly practice gynecological acts.

A lot of studies have studied why general doctors not practice gynecological acts but it would necessary to include the women's perspective.

DETAILED DESCRIPTION:
The aim of the study will be identify women's factors associated with gynaecological consultation by the general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* women aged more than 18 years old
* woman agreeing to participate to the study

Exclusion Criteria:

* women aged less than 18 years old
* woman not agreeing to participate to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women aged more than 18 years old, who consent to participle to the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of gynecological consultation with a general practitioner | Day 0
  would the woman agree to consult a general practitioner for a gynecological reason ? (Yes or No)

SECONDARY OUTCOMES:
Women's knowledge of general practitioner gynecology competences | Day 0
  Does woman know that a general practitioner is able to perform gynecological acts? (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: barbe coralie, Principal Investigator — pratictioner
Locations (1):
- Ufr Medecine Urca, Reims, France

IPD SHARING:
Plan to Share IPD: No